CLINICAL TRIAL: NCT05355012
Title: Organization of Smoking Cessation in Pregnant Women: Study of the Effectiveness, Transferability, Barriers and Facilitators of the Implementation of the 5A Strategy in French Context. A Cluster Randomized Controlled Trial in New Aquitaine.
Brief Title: Organization of Smoking Cessation in Pregnant Women With the Implementation of the 5A Strategy in New Aquitaine.
Acronym: 5A-QUIT-N
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2019/61
Record Dates: First submitted 2022-03-02; First posted 2022-05-02 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Smoking Cessation; Pregnancy Related
Keywords: Smoking cessation; Pregnancy; 5As; Healthcare optimization; Transferability; Healthcare sustainability; Organizational innovation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: In order to evaluate the effectiveness of 5A-QUIT-N, we will conduct a trial in New Aquitaine using a mixed quantitative and qualitative method.
  The quantitative study is a stepped-wedge cluster randomized trial (SWCRT) with a transition phase (deployment). The duration of each period is set at 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5A-QUIT-N intervention (Experimental): The 5A-QUIT-N intervention can be defined as multilevel, i.e., it is based on a territorial organization with expected results at the level of professional practice (structuring of practices around the 5A method) and therefore of the care of pregnant women who smoke tobacco.
  This project is based on three strategic axes:
  * A gradation of the care offer
  * Personalized care by developing specific treatment paths
  * Coordination of territorial resources to support pregnant women in quitting smoking.
  These elements will make it possible to propose a partnership-based, multi-professional, coordinated and integrated approach to the territory, supported by the technical resources and expertise available in the territory. It invites a majority of non-specialized actors to invest in the process of supporting pregnant women in quitting smoking, multiplying and potentiating their actions with this population.
  Interventions: Other: 5A organizational innovation
- 5A-QUIT-N control (No Intervention): Usual care in the care of pregnant women who smoke tobacco.

INTERVENTIONS:
Other: 5A organizational innovation — This project is based on three strategic axes:
  * A gradation of the care offer allowing to adapt the means and resources mobilized on the territory
  * Personalized care by developing specific treatment paths based on the risk factors and/or vulnerabilities of the pregnant woman
  * Coordination of territorial resources to support pregnant women in quitting smoking These three key elements will make it possible to propose a partnership-based, multi-professional, coordinated and integrated approach to the territory, supported by the technical resources and expertise available in the territory. It invites a majority of non-specialized actors to invest in the process of supporting pregnant women in quitting smoking, multiplying and potentiating their actions with this population.
  Arms: 5A-QUIT-N intervention

SUMMARY:
The investigators are conducting a pragmatic cluster randomized trial in stepped-wedge of which objectives are to evaluate the effectiveness and the conditions of effectiveness of an organizational strategy for smoking cessation - 5A-QUIT-N - among pregnant women in New Aquitaine (NA), by using and optimizing existing resources

DETAILED DESCRIPTION:
In France, in 2016, 16.6% of pregnant women were smokers, the highest levels among European countries. Pregnancy is considered a teachable moment for smoking cessation. There are many tools, interventions and programs to reduce the smoking habits of pregnant women. The challenge is therefore not to propose new interventions but to understand what is hindering the implementation of existing interventions and proposing corrective measures. In this context, the scientific literature shows that interventions for smoking pregnant women only seem effective when based on a comprehensive approach that combines multiple interventions. In particular, interventions based on the 5A's model (Ask, Advise, Assess, Assist, Arrange) are largely recommended and have shown their effectiveness abroad. Factors facilitating or hindering the implementation of such strategies are mainly organizational. As organizations are context-dependent by nature, considering the generalization of such strategies in France therefore requires adapting them to the French health system and evaluating them in context, in a pragmatic approach, inserted into routine care and using the tools, procedures and existing organizations in the territories.

ELIGIBILITY:
In this research, there are 4 categories of research participants:

* Healthcare professionals: the target of the 5A-QUIT-N intervention from whom data will be collected to meet the secondary objective of the effectiveness conditions.
* Stakeholders: individuals involved in the implementation of the research and intervention from whom data will be collected to meet the secondary objective of the effectiveness conditions.
* Women who have just given birth and who smoke tobacco in early pregnancy: indirect beneficiaries of the intervention, from whom data will be collected to meet the primary objective of effectiveness.
* Co-parent (partner) of the new-born child of the woman who has just given birth included in the study

Inclusion criteria for the intervention

The inclusion criteria for the clusters are :

- Territory of maternity attractiveness in New Aquitaine

The inclusion criteria for care providers within the clusters are:

* All institutions, structures and organizations and health professionals likely to participate in the follow-up of pregnant women
* All institutions, structures and organizations and health professionals specializing in addictology or tobaccoology

The inclusion criteria for pregnant women within the clusters are :

- All pregnant women who have smoked tobacco (at least 2 times a week, for at least 1 week) during the pregnancy (including the period when she was unaware of the pregnancy)

Inclusion criteria for the primary objective measures:

The inclusion criteria for women are (for data collection):

* Have given birth in a New Aquitaine maternity hospital,
* Reside in New Aquitaine
* To have been followed for the pregnancy in the territory of the maternity of delivery
* To have used tobacco during (at least 2 times a week, for at least 1 week) the pregnancy (including the period when she was unaware of the pregnancy)
* Be over 18
* Have given free, informed and express consent

  * Exclusion criteria:

Non-inclusion criteria for the intervention

Cluster non-inclusion criteria:

* Pilot territory (territory of attractiveness of the Arcachon maternity hospital)
* Impossibility of collecting the main judgment criterion in the cluster Within these clusters, the health care providers and the pregnant women are all concerned and therefore do not have any non-inclusion criteria.

Non-inclusion criteria of measures for the primary objective:

The criteria for non-inclusion of women who have just given birth are:

* Not speaking French,
* Have COVID during delivery
* Use only electronic cigarettes,
* Under legal protection (guardianship, curatorship, safeguard of justice)
* Women giving birth under X
* Women giving birth to a stillborn baby
* Women having made a denial of pregnancy
* Women who have their child in neonatal intensive care
* Women who have been fully monitored for their pregnancy outside of New Aquitaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4505 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Tobacco abstinence at delivery | At delivery (smoking status of the previous 7 days)
  The point prevalence of abstinence at delivery, which is the proportion of women reporting abstinence from smoking for at least 7 days at delivery. This criterion is well documented in the literature assessing tobacco use. It has the advantage of detecting the delayed effects of an intervention and can be easily extrapolated.

SECONDARY OUTCOMES:
Average number of cigarettes smoked at inclusion | At inclusion
  Average number of cigarettes smoked per day over the last 30 (or 7) days
Average number of cigarettes smoked at postpartum | 6 months and 1 year after delivery
  Average number of cigarettes smoked per day over the last 30 (or 7) days
Attempts to reduce tobacco consumption | 1 to 3 days after delivery
  The number of attempts to reduce tobacco consumption (at least 1 cigarette)
Attempts to quit smoking | 1 to 3 days after delivery
  Number of attempts to quit smoking (at least 24 hours)
Continuous abstinence | 1 to 3 days after delivery
  Continuous abstinence (in number of days)
Birth weight | At baby birth, up to 3 days after delivery
  Birth weight (in kg) of the baby
Gestational age | At baby birth, up to 3 days after delivery
  Gestational age (in months) of the baby (at birth).
Sustainability of professional practices | 18 months from the deployment of the intervention
  Prevalence of completion of each A of the 5A approach evaluated on a subgroup of women who have just given birth at a distance from the deployment of the intervention (18 months) via the questionnaire
Sustainability of the impact on health | 18 months from the deployment of the intervention
  Prevalence of women smoking tobacco at delivery over the last 7 days via two sources: the computer systems of the maternity units that have this information systematically (non-exhaustive because not all maternity units in the New Aquitaine region have a computer system) and on a sub-group of women who have just given birth
Postpartum relapse rate at 6 months | At 6 months postpartum
  Relapse rate among women who quit smoking during pregnancy at 6 and 12 months postpartum defined as a resumption of at least 7 consecutive days of smoking in the past 6 months.
Postpartum relapse rate at 12 months | At 12 months postpartum
  Relapse rate among women who quit smoking during pregnancy at 6 and 12 months postpartum defined as a resumption of at least 7 consecutive days of smoking in the past 6 months.
Continued abstinence | 6 months and 1 year after delivery
  Continued abstinence (in number of days)
Implementation of intervention | Through study completion, an average of 3 years
  Barriers and levers to implementation in professionals
Conditions of transferability | Through study completion, an average of 3 years
  Conditions of transferability linked to the characteristics of the stakeholders and the context: contextual conditions for success within the centres, the characteristics of professionals and patients influencing outcomes
Viability | Through study completion, an average of 3 years
  Assessment of intervention deployment in a real-world setting, using 5 criteria: utility, affordability, evaluability, adaptability and acceptability.
  "Utility" dimension (as a complement to the secondary criteria) of viability through the recovery mechanisms identified as successful mental health recovery Affordability for professionals and beneficiaries (financial, geographical, social and cultural levers and brakes of the intervention) Evaluability of 5A-QUIT-N: carrying out this evaluation, the availability of professionals and beneficiaries to answer questionnaires and interviews, missing data in the questionnaires etc.
  Adaptability of 5A-QUIT-N: integration of the action into the context and the current organisation of the centres Acceptability of 5A-QUIT-N: by professionals and beneficiaries

CONTACTS AND LOCATIONS:
Overall Officials: François Alla, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Hôpital Saint-André, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No